CLINICAL TRIAL: NCT04076982
Title: Effect of Supplementary Dietary Protein (21g Per Day) on Lean Mass and Strength in Sedentary, Adult Vegetarians
Acronym: MungBean
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: Christopher Wharton (Unknown); Eric Bartholomae (Unknown); April Incollingo (Unknown); Maricarmen Vizcaino (Unknown)
Responsible Party: Principal Investigator, Carol Johnston, Professor and Associate Dean, Arizona State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: MungBean00005383
Record Dates: First submitted 2019-08-29; First posted 2019-09-04 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-09

CONDITIONS: Muscle Weakness
Keywords: vegetarian; vegan; plant-based; protein; strength
MeSH Terms: conditions — Muscle Weakness

STUDY DESIGN:
Intervention Model Description: Qualifying participants will be stratified and randomly assigned to one of two treatment arms: mung bean protein or control biscuit. Participants will meet with study investigators on two occasions separated by 8 weeks for assessments.
Who Masked: Participant
Masking Description: Participants were told that the study investigated the impact of a dietary intervention on body composition and strength. The 'egg patty' and 'biscuit' were referred to as dietary supplements.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mung bean (Experimental): daily oral administration of protein supplement
  Interventions: Dietary Supplement: mung bean protein
- biscuit (Placebo Comparator): daily oral administration of control supplement
  Interventions: Other: control biscuit

INTERVENTIONS:
Dietary Supplement: mung bean protein — Participants were instructed to consume the test foods in the morning hours and to keep a record of the days the foods were consumed on a study calendar which was returned to investigators at the final visit and used to track protocol adherence.
  Arms: mung bean
Other: control biscuit — Participants were instructed to consume the test foods in the morning hours and to keep a record of the days the foods were consumed on a study calendar which was returned to investigators at the final visit and used to track protocol adherence.
  Arms: biscuit

SUMMARY:
It is possible that the lower protein intake in vegetarians and vegans may relate to a decrease in grip strength. Furthermore, there is limited research examining the effects of plant-based protein intake on strength and LBM independent of an exercise training component. The present study was designed to examine relationships between strength, protein intake, and LBM in underactive vegetarian and vegan adults, as well as the impact of protein supplementation (18 g mung bean protein daily) on these indices.

DETAILED DESCRIPTION:
The American Dietetic Association states that based off of evidence, it is possible for a vegetarian to obtain the recommended amount of nutrients with a properly planned diet. By mixing various sources of plant proteins throughout the day, a person can obtain all the amino acids needed for growth and tissue maintenance and repair. Yet, many vegetarians struggle to eat a substantial diet, especially when it comes to protein. This is because plant protein has protein bioavailability that is 10-30% lower than animal protein. As a result, current research suggests that there needs to be a separate protein dietary reference intake (DRI) for vegetarians and it needs to be larger than the protein DRI for omnivores. Whenever considering protein bioavailability, the quality must be assessed by analyzing the digestibility, chemical integrity, and freedom from interference in metabolism of the amino acid. This is a major concern because inadequate protein intake can affect bone health and alter muscle mass. Importantly, research has shown as a result of inadequate protein intake, vegetarians tend to have less lean body mass and less muscle strength than omnivores. Currently, all research available on this topic included strength training as a variable for increasing lean muscle mass, and no research has been reported that analyzed the impact of increased dietary protein on lean body mass without a training component. This parallel arm study will examine the effect of supplemental plant protein on strength and lean body mass in adult, non-athletic vegetarians in the Phoenix area.

ELIGIBILITY:
Inclusion Criteria:

* vegetarian or vegan for at least one year
* healthy by self-report

Exclusion Criteria:

* supplement use such as protein powder or creatine
* previous diagnosis of heart disease, cancer, stroke, diabetes, autoimmune disorders, or thyroid condition
* competition in any athletic event in the past year
* moderate to strenuous exercise exceeding 150 minutes per week
* pregnant or planning to become pregnant.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2018-09-03 (Actual); Primary Completion 2019-01-12 (Actual); Study Completion 2019-01-12 (Actual)

PRIMARY OUTCOMES:
grip strength | change in strength from baseline to week 8
  Dominant handgrip strength was measured in triplicate in a seated position with the elbow flexed to 90 degrees and a neutral wrist position in triplicate using a handheld dynamometer
leg strength | change in strength from baseline to week 8
  Lower body strength was measured in the dominant leg using a multi-joint system dynamometer. Isokinetic knee flexion and extension were measured from a seated position at a resistance of 90°/sec.

SECONDARY OUTCOMES:
lean body mass | change in LBM from baseline to week 8
  LBM was measured via dual energy X-ray absorptiometry (DEXA) and was conducted by a trained X-ray technician.

CONTACTS AND LOCATIONS:
Locations (1):
- Arizona State University, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No